CLINICAL TRIAL: NCT02785393
Title: Doxazosin as a Potential Treatment for Methamphetamine Dependence
Brief Title: DOX as a Potential Treatment for Methamphetamine Dependence
Acronym: DOX-Meth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas Newton, Professor, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H-26957; DPMC (Other: NIDA); P50DA018197 (NIH)
Record Dates: First submitted 2014-09-24; First posted 2016-05-27 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Substance-Related Disorders
Keywords: Methamphetamine; Dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Sugars; Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill
- Doxazosin (Active Comparator)
  Interventions: Drug: Doxazosin

INTERVENTIONS:
Drug: Sugar Pill — The administration of a sugar pill
  Arms: Sugar Pill
Drug: Doxazosin — The administration of the Doxazosin medication
  Arms: Doxazosin

SUMMARY:
The purpose of the study is to asses the potential interactions between methamphetamine and doxazosin in methamphetamine-dependent volunteers who are not seeking treatment. The study will evaluate the effects of doxazosin on the cardiovascular and subjective effects of methamphetamine in a human laboratory study.

The primary objective is to determine the safety of treatment with doxazosin in methamphetamine-dependent volunteers by examining hemodynamic and subjective effects of administration of ascending doses of methamphetamine and a placebo dose during treatment with doxazosin.

The secondary objective is to determine effects of treatment with doxazosin, as compared to placebo, on subjective effects produced by administration of methamphetamine or placebo

DETAILED DESCRIPTION:
Purpose:

To determine the effects of treatment with doxazosin, compared to treatment with placebo, on methamphetamine-induced craving and subjective effects in methamphetamine-dependent human volunteers.

Secondary aims are to clarify the genetics of substance abuse, potentially leading to improved methods to diagnosis those at risk and to help develop better therapeutic interventions and to develop a new saliva-based test for the detection and measurement of drugs of abuse.

Design/Procedure:

Twenty non-treatment-seeking methamphetamine-dependent volunteers will complete procedures during treatment with placebo and study medication, in random order, using a within-subjects, double-blind, placebo-controlled design. There will be a two week period between each phase. The dose of doxazosin needed to alter the effects of methamphetamine is unknown and preclinical animal studies have not been conducted. Because of this, initially the investigators will study the effects of a low dose of doxazosin (4mg daily) compared to placebo daily. Methamphetamine (0, 10, and 30mg, smoked) will be administered during treatment with 4mg doxazosin/placebo. Methamphetamine will be administered in ascending dose (10mg followed by 20mg) with the 0mg dose randomly interspersed to maintain the blind. Cardiovascular measures and subjective effects ratings will be assessed following methamphetamine administration.

Participants will be monitored for stability on days 11 and 12 and discharged from the hospital on day 13.

If 4mg doxazosin treatment is well tolerated but is not associated with alterations in the effects of methamphetamine, a second group of subjects will be studied using the same sample size. Treatment will begin at 1mg and increased by 1mg increments every three days until 8mg is reached. Placebo will be dosed identically. All study procedures will be identical as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Be English-speaking volunteers who are not seeking treatment at the time of the study
2. Be between 18-55 years of age
3. Meet DSM-IV TR criteria for methamphetamine dependence; participants may or may not meet criteria for nicotine dependence. Nicotine dependence is allowed but not required because most methamphetamine users smoke cigarettes.
4. Have a self-reported history of using methamphetamine by the smoked or IV route
5. Have vital signs as follows: supine blood pressure > 100/65 mm Hg, a seated blood pressure of > 90/60 mm Hg, and an orthostatic change < 20 mm Hg systolic or <10 mm Hg diastolic on standing. To ensure that subjects will not be at risk from methamphetamine, the resting pulse must be < 90 bpm and the blood pressure must be < 150 mmHg systolic and < 90 mmHg diastolic.
6. Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) within normal limits
7. Have a baseline EKG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant arrhythmias
8. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.

Exclusion Criteria:

1. Meet DSM IV TR criteria for dependence on drugs other than methamphetamine or nicotine.
2. Have any history or evidence suggestive of seizure disorder or brain injury
3. Have any previous medically adverse reaction to methamphetamine, including loss of consciousness, chest pain, or epileptic seizure
4. Have neurological or psychiatric disorders, such as:

   * psychosis, bipolar illness or major depression as assessed by MINI
   * organic brain disease or dementia assessed by clinical interview
   * history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult
   * history of suicide attempts within the past year and/or current suicidal ideation/plan
5. Have evidence of clinically significant heart disease or hypertension, as determined by the PI
6. Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
7. Have symptomatic HIV or are taking antiretroviral medication
8. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation
9. Have asthma or currently use theophylline or other sympathomimetics
10. Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Criteria for Discontinuation Following Initiation Participants will be discharged if they have a positive breath test indicating use of alcohol or a urine test indicating illicit use of drugs while in the MED-VAMC, if they do not comply with study procedures, or if they do not tolerate the study drugs. Stopping criteria are detailed below.

Subject Selection Criteria Rationale Route of administration. Participants are required to have used MA by the IV or smoked route to avoid exposing participants to drugs by routes of administration that produce more intensive interoceptive effects than usually used by the participants. Prior experience with smoked MA is allowed (rather than restricting the population to those with experience with IV MA) because smoked MA reaches brain sites of action as rapidly as does intravenously administered MA and smoked MA produces effects that are comparable to IV MA. Speed of administration (and rate of delivery to brain) of stimulant drugs likely impacts subjective and cardiovascular effects, so smoked and intravenously administered MA produce similar subjective effects (22-26).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
blood pressure, change from baseline | -15 min, 15 min, 30 min, 45 min, 60 min post-MA dosing
heart rate, change from baseline | -15 min, 15 min, 30 min, 45 min, 60 min post-MA dosing

SECONDARY OUTCOMES:
subjective effects of methamphetamine or placebo, change from baseline | -15 min, 5 min, 15 min, 30 min, 45 min and 60 min after MA dosing
  Subjective effects are drug effects including euphoria, desire, anxiety, stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Newton, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael Debakey VA Medical Center, Houston, Texas, United States